CLINICAL TRIAL: NCT02652481
Title: Expanding MRI (Magnetic Resonance Imaging) Access for Patients With New and Existing ICDs (Implantable Cardioverter Defibrillator) and CRT-Ds (Cardiac Resynchronization Therapy Defibrillator)
Brief Title: ENABLE MRI (Magnetic Resonance Imaging)
Acronym: ENABLE-MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: C1734
Record Dates: First submitted 2016-01-08; First posted 2016-01-12 (Estimated); Results first posted 2019-07-16 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- ImageReady MR Conditional Defibrillation System Group (Other): Prospective, non-randomized, confirmatory study.Subjects will initially be enrolled into Phase I to undergo a non-diagnostic study required MR Scan. Once Phase I is complete, subjects will be enrolled into Phase II where there is no requirement to undergo a non-diagnostic study required MR scan Up to 37 subjects will be used for an interim analysis. Of these subjects, the first 20 who undergo the study required MRI scan and complete the MRI + 1 Month Visit will be used for this analysis. The second cohort will consist of subjects who will receive the non-diagnostic study required MR scan until 137 CRT-D and 28 VR ( single chamber) ICD subjects undergo the study required MR scan (complete or incomplete).
  De novo implants and existing implants may be enrolled in Phase I There will be a non-diagnostic study required MR scan (during the MRI visit) There will be a study required MRI visit and MRI + 1 month visit
  Interventions: Device: ImageReady MR Conditional Defibrillation System

INTERVENTIONS:
Device: ImageReady MR Conditional Defibrillation System — ImageReady MR Conditional Defibrillation System Components:
  Device Name Device Model Number Pulse Generators Phase I and II Phase II Only * CRT-D (IS1/DF4/IS4) VR ICD (DF4) DR ( dual chamber) ICD (IS1/DF4) ORIGEN™ MINI ICD ORIGEN EL ICD ORIGEN X4 CRT INOGEN™ MINI ICD INOGEN EL ICD INOGEN X4 CRT DYNAGEN™ MINI ICD DYNAGEN EL ICD DYNAGEN X4 CRT-D AUTOGEN ™ MINI ICD* AUTOGEN EL ICD* AUTOGEN X4 CRT-D* Right Atrial Leads and Accessories FINELINE™ II Sterox FINELINE II Sterox EZ Suture Sleeves for FINELINE II Leads INGEVITY™ MRI* Suture Sleeve for INGEVITY MRI* IS-1 Lead Port Plug 7145 Right Ventricular Leads and Accessories RELIANCE 4-FRONT™ (DF4)* Suture Sleeve for RELIANCE 4-FRONT leads*; ENDOTAK RELIANCE™ (DF4) Left Ventricular Leads and Accessories ACUITY™ X4 (IS4) Suture Sleeve for ACUITY X4 leads
  * May only be used internationally outside the US

SUMMARY:
The objective of this study is to collect data to confirm the safety and effectiveness of the Image Ready™ MR (Magnetic Resonance) Conditional Defibrillation System when used in the 1.5T (Tesla) MRI environment under the labeled Conditions of Use (Phase I).

Additionally, the study will assess medically necessary MR scans according to the labeled Conditions of Use to provide real-world scanning data (Phase I and Phase II).The study also aims to demonstrate the continued ability of the ImageReady MR Conditional Defibrillation System to sense and detect ventricular fibrillation (VF) post MRI scan by collecting and analyzing data from spontaneous VF episodes, "for-cause" VF inductions, and from an optional VF induction Sub-study.

.

ELIGIBILITY:
Key Inclusion Criteria:

1. Phase I: Subject is indicated per guidelines and will receive a CRT-D or ICD system OR Subject is implanted with a functional and stable CRT-D or ICD system Phase II: Subject is implanted with a functional and stable CRT-D or ICD system
2. Subject will receive or is implanted with an ICD or CRT-D pulse generator in the left or right pectoral region
3. Subject is able and willing to undergo an MR scan without intravenous sedation (Phase I only)
4. Subject is willing and capable of providing informed consent and participating in all testing/ visits associated with this clinical study at an approved clinical study center and at the intervals defined by this protocol
5. Subject is age 18 or above, or of legal age to give informed consent specific to state and national law

Key Exclusion Criteria:

1. Subject implanted with an ICD or CRT-D pulse generator with battery at Explant status
2. Subject has other active or abandoned implanted cardiac rhythm devices, components or accessories present such as pulse generators, leads, lead adaptors or extenders
3. Presence of metallic objects that represent a contraindication to MR imaging at the discretion of the Radiologist and impacting the ability to conduct the study protocol
4. Subject needs or will need a medically necessary MR scan, before completing the 1-month post-MR follow-up visit (Phase I only)
5. Subject with:

   * A history of syncope related to brady-arrhythmia
   * A history of syncope of unknown etiology
   * Sinus pauses (Pause > 2 s)
   * Permanent or intermittent complete AV (Atrioventricular ) block
   * Documentation of progressive AV nodal block over time
   * Trifascicular block (alternating bundle branch block or PR > 200 ms (interval between P wave and R-wave) with LBBB ( Left bundle branch block) or other bifascicular block) Note: It is required to run a 12 lead ECG (Electrocardiography) and a 10s rhythm strip to document this exclusion criterion. During ECG acquisition, subjects must be in either their own intrinsic rhythm or, in subjects with an existing device implant, the device must be programmed to VVI (ventricular demand pacing) 40 ppm.
6. Subject is not clinically capable of tolerating the absence of pacing or Resynchronization therapy support in a supine position for the duration that the pulse generator is in MRI Protection Mode, per Physician discretion
7. Subject is not clinically capable of tolerating the absence of Tachycardia therapy support for the duration that the pulse generator is in MRI Protection Mode, per Physician discretion
8. Subjects with a planned RA( right atrium), RV ( right ventricle) or LV (left ventricle) lead revision or extraction within 30 days of enrollment (Phase I only)
9. Subjects with an implanted lead that is planned to be extracted during the study implant procedure
10. Subjects currently requiring dialysis
11. Subject has a mechanical heart valve
12. Subject has a known or suspected sensitivity to dexamethasone acetate (DXA)
13. Subject is currently on the active heart transplant list
14. Subject has documented life expectancy of less than 12 months
15. Subject is enrolled in a concurrent study, with the exception of local mandatory governmental registries and observational studies/registries, without the written approval from Boston Scientific
16. Women of childbearing potential who are or might be pregnant, and will receive an ICD or CRT-D pulse generator

VF Induction Sub-study Exclusion Criteria:

In addition to meeting all of the inclusion criteria and none of the exclusion criteria of the ENABLE MRI study, subjects enrolled in the VF Induction Sub-study must also not meet any of the following VF Induction Sub-study exclusion criteria:

1. Unstable heart failure requiring hospitalization in the last 30 calendar days
2. Unable to tolerate sedation (e.g. IV (intravenous sedation )sedation, general anesthesia)
3. Planned cardiac revascularization procedure
4. Right Ventricular Lead R wave is less than 5 mV(milliVolt)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2016-01; Primary Completion 2017-04-30 (Actual); Study Completion 2018-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Voss, Study Director — Boston Scientific Corporation
Locations (57):
- United States (34):
  - Heart Center Research, LLC, Huntsville, Alabama
  - Cardiology Associates of Northeast Arkansas, Jonesboro, Arkansas
  - Huntington Memorial Hospital, Pasadena, California
  - University of California - San Diego-N, San Diego, California
  - John Muir Medical Center, Walnut Creek, California
  - Manatee Memorial Hospital, Bradenton, Florida
  - Lakeland Regional Medical Center, Lakeland, Florida
  - University Community Hospital, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - St. John's hospital, Springfield, Illinois
  - St. Vincent's Hospital, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Marquette General Hospital, Marquette, Michigan
  - Centracare Heart and Vascular Center, Saint Cloud, Minnesota
  - HealthEast St. Joseph's Hospital, Saint Paul, Minnesota
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Cox Health, Springfield, Missouri
  - Northwell Health, New York, New York
  - University of North Carolina Hospital, Chapel Hill, North Carolina
  - OhioHealth Research and Innovation Institute - Riverside Methodist Hospital, Columbus, Ohio
  - The Toledo Hospital, Toledo, Ohio
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Bryn Mawr Medical Specialists, Bryn Mawr, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - St. Thomas Research Institute, LLC, Nashville, Tennessee
  - SouthEast Texas Clinical Research Center, Beaumont, Texas
  - University of Texas Houston Health Science Center, The Woodlands, Texas
  - Trinity Mother Frances Health System, Tyler, Texas
  - University of Utah Hospital and Clinics, Salt Lake City, Utah
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Virginia Commonwealth University Health System, Richmond, Virginia
  - Providence Regional Medical Center Everett, Everett, Washington
  - PeaceHealth Southwest Medical, Vancouver, Washington
- Academisch Ziekenhuis Middelheim, Antwerp, Belgium
- Germany (3):
  - Deutsches Herzzentrum Berlin, Berlin
  - Medizinische Hochschule Hannover MHH, Hanover
  - Klinikum Magdeburg, Magdeburg
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Israel (4):
  - Rambam Medical Center, Haifa
  - Soroka MC, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Hadassah Hebrew University Medical Center, Tel Litwinsky
- Italy (7):
  - Fondazione di Ricerca e Cura 'Giovanni Paolo II', Campobasso
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Ospedaliera San Camillo-Forlanini, Roma
  - Ospedale S.G. Calibita Fatebenefratelli - Isola Tiberina, Roma
  - Ospedale san giovanni calibita, Roma
  - Policlinico Casilino, Roma
  - Osp. S. Maria Della Misericordia, Udine
- Malaysia (2):
  - Institut Jantung Negara, Kuala Lumpur
  - University of Malaya Medical Centre, Kuala Lumpur
- Hospital Clinic de Barcelona, Barcelona, Spain
- United Kingdom (3):
  - Heart and Chest Hospital, Liverpool
  - Guys and St. Thomas NHS Foundation Trust, London
  - Freeman Hospital, Newcastle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rinaldi CA, Vitoff PJ, Nair DG, Bernstein R, Mountantonakis SE, Rapacciuolo A, Carter N, Tse HF, Green UB. Safety of magnetic resonance imaging scanning in patients with cardiac resynchronization therapy-defibrillators incorporating quadripolar left ventricular leads. Heart Rhythm. 2020 Dec;17(12):2064-2071. doi: 10.1016/j.hrthm.2020.08.020. Epub 2020 Sep 7. PMID 32911050

RESULTS

PARTICIPANT FLOW:
Groups:
- ImageReady MR Conditional Defibrillation System Group: This is a prospective, non-randomized, confirmatory study. Some defibrillator systems are not able to be used with MRI scanners because the material they are made out. Boston Scientific has a defibrillation system with a new feature that blocks interference from an MRI scanner when the defibrillator system is set to the "MRI protection mode". This new MRI scan feature was considered "investigational" , meaning was investigated because it was not approved by the US Food and Drug Administration (FDA) for patient use. This new defibrillation system is called the ImageReady Defibrillation System. Together, the defibrillator and the lead(s) are called the ImageReady System. The ImageReady system is considered investigational in the US because not all the component parts are approved by the FDA. Patients who have a ImageReady defibrillator will undergo an MRI and data will be collected. Periodic checks were planned to check the defibrillator system.
Period: Phase 1
Arm/Group | ImageReady MR Conditional Defibrillation System Group
Started | 239
Completed | 141
Not Completed | 98
Period: Phase 2
Arm/Group | ImageReady MR Conditional Defibrillation System Group
Started | 261
Completed | 243
Not Completed | 18

BASELINE CHARACTERISTICS:
Population: Subjects enrolled into Phase I and underwent a required (non-diagnostic, non-medically necessary) MRI. The data from phase I (N=237) was used for the PMA application and approval. Enrollment was stopped for phase II once 500 enrolled subjects were reached. Baseline participants are 498 patients as two patients were enrolled in error.
Groups:
- ImageReady™ MR Conditional Defibrillation System: This is a prospective, non-randomized, confirmatory study. Some defibrillator systems are not able to be used with MRI scanners because the material they are made out. Boston Scientific has a defibrillation system with a new feature that blocks interference from an MRI scanner when the defibrillator system is set to the "MRI protection mode". This new MRI scan feature was considered "investigational" , meaning was investigated because it was not approved by the US Food and Drug Administration (FDA) for patient use. This new defibrillation system is called the ImageReady Defibrillation System. Together, the defibrillator and the lead(s) are called the ImageReady System. The ImageReady system is considered investigational in the US because not all the component parts are approved by the FDA. Patients who have a ImageReady defibrillator will undergo an MRI and data will be collected. Periodic checks were planned to check the defibrillator system.
Arm/Group | ImageReady™ MR Conditional Defibrillation System
Number analyzed (Participants) | 498
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136
  Male | 362
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 381
  Race: Black or African heritage | 45
  Race: Hispanic or Latino | 6
  Race: Asian | 42
  Race: Other | 5
  Race: American Indian | 3
  Race: Unknown | 16
Region of Enrollment [Count of Participants; unit: Participants]
  Hong Kong | 19
  Belgium | 3
  United States | 302
  Italy | 87
  United Kingdom | 20
  Malaysia | 20
  Israel | 6
  Germany | 19
  Spain | 10
  Austria | 12
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.0 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Free From MR (Magnetic Resonance) Scan-related Complications
Description: MR scan-related CFR (Complication-free rate) between the MR Scan and the MRI + 1 (Magnetic Resonance Imaging) Month Visit
Time Frame: The time between the MR Scan and MRI + 1 Month
Population: All implanted subjects that completed any portion of the study required MR scan and did not have a Medically Necessary Scan (MNS) performed prior to the MRI+1 Month Visit were included in the Primary Safety Endpoint analysis set.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | ImageReady MR Conditional Defibrillation System Group
Number analyzed (Participants) | 159
percentage of participants | 100 [100 to 100]

2. Primary Outcome: Percentage of Participants That Had an Increase in Average Pacing Thresholds ≤ 0.5V (Volt) (at 0.5 ms) in the RV
Description: Increases in RV pacing threshold (at 0.5 ms) pre- MR scan and 1 Month post-MR scan were calculated for subjects. Subjects that had an increase in average pacing thresholds ≤ 0.5V (at 0.5 ms) from pre-MR Scan to MRI Visit + 1 Month follow-up were considered a success.
Time Frame: The time between the MR Scan and MRI + 1 Month
Population: Did not include subjects that had a MNS between implant and the MRI+1Month Visit; Failed to meet Conditions of Use; Experienced lead-related complication; Had an incomplete scan or no scan, died or withdrew consent, missed a visit, missed lead measurements
Measure: Number (95% Confidence Interval); unit: percentage of participants with success
Arm/Group | ImageReady MR Conditional Defibrillation System Group
Number analyzed (Participants) | 146
percentage of participants with success | 99.32 [96.79 to 100]

3. Primary Outcome: Percentage of Participants That Had an Increase in Average LV ( Left Ventricle) Pacing Threshold ≤ 1.0V (Volt) at 0.5 ms.
Description: Increases in average LV pacing threshold (at 0.5 ms) pre- MR scan and 1 Month post-MR scan were calculated for subjects. Subjects that had an increase in pacing thresholds measurements ≤ 1.0V (at 0.5 ms) from pre-MR Scan at MRI Visit to MRI + 1 Month Visit were considered a success.
Time Frame: The time between the MR Scan and MRI + 1 Month
Population: did not include subjects with a MNS between implant and the MRI + 1 Month Visit;failed to meet labeled MRI Conditions of Use, had lead-related complication;had an incomplete scan or no scan; missing lead measurements; missed a visits, subject died or withdrew consent
Measure: Number (95% Confidence Interval); unit: percentage of participants with succes
Arm/Group | ImageReady MR Conditional Defibrillation System Group
Number analyzed (Participants) | 120
percentage of participants with succes | 100 [97.53 to 100]

4. Primary Outcome: Percentage of Participants That Had a Decrease in RV ( Right Ventricle) Sensed Amplitude
Description: Decreases in RV sensed amplitude pre-MR scan and 1 Month post-MR scan were calculated for subjects. Subjects were considered a success if the average sensed amplitude at the MRI + 1 Month Visit remains ≥ 5.0 mV and above 50% of the pre-MR scan value. Subjects who had an average pre-scan RV sensed amplitude measurement < 5.0 mV were excluded from this analysis.
Time Frame: The time between the MR Scan and MRI + 1 Month
Population: Did not include subjects that had a MNS between implant and the MRI+1Month Visit; Failed to meet Conditions of Use; Experienced lead-related complication; Had an incomplete scan or no scan, died or withdrew consent, missed a visit, missed lead measurements; had an average pre-scan RV sensed amplitude measurement < 5.0 mV.
Measure: Number (95% Confidence Interval); unit: percentage of participants with succes
Arm/Group | ImageReady MR Conditional Defibrillation System Group
Number analyzed (Participants) | 146
percentage of participants with succes | 99.32 [96.79 to 100]

5. Primary Outcome: Percentage of Participants That Decrease in LV ( Left Ventricle) Sensed Amplitude
Description: Decreases in average LV sensed amplitude pre-MR scan and 1 Month post-MR scan were calculated for subjects. Subjects were considered a success if the average sensed amplitude at the MRI + 1 Month Visit remained ≥ 5.0 mV and above 50% of the average pre-MR scan value. Subjects who had an average pre-scan LV sensed amplitude measurement < 5.0 mV were excluded from this analysis.
Time Frame: The time between the MR Scan and MRI + 1 Month
Population: did not include subjects with a MNS between implant and the MRI + 1 Month Visit;failed to meet labeled MRI Conditions of Use, had lead-related complication;had an incomplete scan or no scan; missing lead measurements; missed a visits, subject died or withdrew consent; Average LV sensed amplitude <5mV (3 patients)
Measure: Number (95% Confidence Interval); unit: percentage of participants with succes
Arm/Group | ImageReady MR Conditional Defibrillation System Group
Number analyzed (Participants) | 118
percentage of participants with succes | 98.31 [94.76 to 100]

ADVERSE EVENTS:
Time Frame: Safety data are presented for subjects as from enrollment until study completion ( 4 May 2018)
Description: Investigators were asked to classify whether an adverse event was considered serious or nonserious,whether it was anticipated or unanticipated; met USADE(Unanticipated Serious Adverse Device Effect); UADE (Unanticipated Adverse Device Effect) definition and whether it was device or procedure related. All reportable events experienced by the study subject after giving informed consent were to be reported. Two patients were enrolled in error and three patients were withdrawn (intent); 495 at risk
Arm/Group | ImageReady MR Conditional Defibrillation System Group
All-Cause Mortality (participants affected / at risk) | 18/495
Serious Adverse Events (participants affected / at risk) | 139/495
Other Adverse Events (participants affected / at risk) | 122/495
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ImageReady MR Conditional Defibrillation System Group (N=495)
Unable to capture - LV PG System (Product Issues) | 0 (0)
Extracardiac stimulation - LV PG System (Product Issues) | 0 (0)
Inappropriate Tachy Therapy - SVT - PG System Therapy (Product Issues) | 1 (1)
Pacemaker Mediated Tachycardia - PG System Therapy (Product Issues) | 0 (0)
Infection (>30 days post-implant) - PG System - Subject related (Infections and infestations) | 6 (6)
Dislodgment - Elevated threshold -RV Lead (Product Issues) | 1 (1)
Dislodgment - Multiple signs - RV Lead (Product Issues) | 1 (1)
Dislodgment - No reported signs - RV Lead (Product Issues) | 2 (2)
Dislodgment - No reported signs - LV Lead (Product Issues) | 1 (1)
Post-surgical wound discomfort/bruising/swelling (Injury, poisoning and procedural complications) | 0 (0)
Adverse reaction - Respiratory - Procedure (Injury, poisoning and procedural complications) | 1 (1)
Hematoma - Pocket (<=30 days post-implant) (Injury, poisoning and procedural complications) | 0 (0)
Pneumothorax - Procedure (Injury, poisoning and procedural complications) | 2 (2)
Pericardial effusion - Procedure (Injury, poisoning and procedural complications) | 0 (0)
Venous occlusion - Procedure (Injury, poisoning and procedural complications) | 0 (0)
Other - PG system procedure (Injury, poisoning and procedural complications) | 1 (1)
Dyspnea - Heart failure (Cardiac disorders) | 8 (9)
Peripheral edema - Heart failure (Cardiac disorders) | 4 (4)
Hypotension - Heart failure (Cardiac disorders) | 0 (0)
Heart failure symptoms - Unspecified (Cardiac disorders) | 11 (11)
Multiple heart failure symptoms (Cardiac disorders) | 28 (37)
Ventricular Fibrillation (VF) (Cardiac disorders) | 4 (5)
Ventricular Tachycardia (VT)/Monomorphic VT (Cardiac disorders) | 5 (6)
Nonsustained Ventricular Tachycardia (NSVT) (Cardiac disorders) | 0 (0)
Atrial Fibrillation (AF) (Cardiac disorders) | 5 (6)
Sinus tachycardia (Cardiac disorders) | 0 (0)
Atrial Tachycardia/Other SVT (eg AVRT, AVNRT, EAT) (Cardiac disorders) | 2 (2)
Atrial (Type I) Flutter (Cardiac disorders) | 2 (2)
Hypotension/Orthostatic Hypotension (Cardiac disorders) | 1 (1)
Hypertension/Hypertensive Crisis (Cardiac disorders) | 1 (2)
Cardiogenic shock (Cardiac disorders) | 2 (2)
Cardiac arrest (Cardiac disorders) | 3 (3)
Myocardial infarction (Cardiac disorders) | 4 (4)
Coronary Artery Disease (Cardiac disorders) | 5 (5)
Peripheral vascular disease (Cardiac disorders) | 6 (6)
Syncope (Cardiac disorders) | 1 (1)
Dizziness (Cardiac disorders) | 0 (0)
Chest pain - Ischemic (Cardiac disorders) | 4 (4)
Chest pain - Other (Cardiac disorders) | 4 (4)
Palpitations (Cardiac disorders) | 0 (0)
Adverse reaction - Hypotension (Vascular disorders) | 0 (0)
Adverse reaction - Anesthesia (Injury, poisoning and procedural complications) | 1 (1)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 8 (15)
Adverse reaction - Medication (Injury, poisoning and procedural complications) | 2 (2)
Systemic infection (Blood and lymphatic system disorders) | 10 (11)
Physical trauma (Skin and subcutaneous tissue disorders) | 1 (1)
Abnormal laboratory values (Blood and lymphatic system disorders) | 0 (0)
Localized Infection (Skin and subcutaneous tissue disorders) | 2 (2)
Neurological (Nervous system disorders) | 3 (3)
Gastrointestinal (Gastrointestinal disorders) | 13 (20)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 17 (19)
Genitourinary (Reproductive system and breast disorders) | 5 (6)
Renal (Renal and urinary disorders) | 7 (8)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 9 (11)
Psychological (Psychiatric disorders) | 1 (2)
Endocrine (Endocrine disorders) | 10 (12)
Cancer (General disorders) | 7 (9)
Multi-system failure (General disorders) | 3 (3)
Unable to capture - RV Lead (Product Issues) | 1 (1)
Conductor coil fracture - RA Lead (Product Issues) | 1 (1)
Migration - PG System - Subject related (Product Issues) | 1 (1)
Myocardial perforation with tamponade (Cardiac disorders) | 1 (1)
Chest pain - Heart failure (Cardiac disorders) | 2 (2)
Pulmonary edema - Heart failure (Cardiac disorders) | 3 (3)
Renal insufficiency/failure - Heart failure (Cardiac disorders) | 3 (3)
Dehydration - Heart failure (Cardiac disorders) | 1 (1)
Gastrointestinal - Heart failure (Cardiac disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1)
Mitral regurgitation (Cardiac disorders) | 1 (1)
Valvular damage/Valvular insufficiency (Cardiac disorders) | 1 (1)
Transient Ischemic Attack (TIA) (Cardiac disorders) | 1 (1)
Cerebrovascular Accident (CVA) (Cardiac disorders) | 4 (4)
Intracardiac thrombus (Cardiac disorders) | 1 (1)
Incessant VT/VT Storm (Cardiac disorders) | 2 (2)
Fever and/or Virus (Infections and infestations) | 2 (2)
Hematological (Blood and lymphatic system disorders) | 3 (3)
Integumentary (Skin and subcutaneous tissue disorders) | 3 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ImageReady MR Conditional Defibrillation System Group (N=495)
Unable to capture - LV PG System (Product Issues) | 2 (2)
Extracardiac stimulation - LV PG System (Product Issues) | 20 (20)
Inappropriate Tachy Therapy - SVT - PG System Therapy (Product Issues) | 6 (6)
Pacemaker Mediated Tachycardia - PG System Therapy (Product Issues) | 4 (4)
Infection (>30 days post-implant) - PG System - Subject related (Infections and infestations) | 2 (2)
Dislodgment - Elevated threshold -RV Lead (Product Issues) | 0 (0)
Dislodgment - Multiple signs - RV Lead (Product Issues) | 0 (0)
Dislodgment - No reported signs - RV Lead (Product Issues) | 0 (0)
Dislodgment - No reported signs - LV Lead (Product Issues) | 0 (0)
Post-surgical wound discomfort/bruising/swelling (Injury, poisoning and procedural complications) | 3 (3)
Adverse reaction - Respiratory - Procedure (Injury, poisoning and procedural complications) | 1 (1)
Hematoma - Pocket (<=30 days post-implant) (Injury, poisoning and procedural complications) | 4 (4)
Pneumothorax - Procedure (Injury, poisoning and procedural complications) | 0 (0)
Pericardial effusion - Procedure (Injury, poisoning and procedural complications) | 1 (1)
Venous occlusion - Procedure (Injury, poisoning and procedural complications) | 1 (1)
Other - PG system procedure (Injury, poisoning and procedural complications) | 0 (0)
Dyspnea - Heart failure (Cardiac disorders) | 4 (4)
Peripheral edema - Heart failure (Cardiac disorders) | 4 (4)
Hypotension - Heart failure (Cardiac disorders) | 1 (1)
Heart failure symptoms - Unspecified (Cardiac disorders) | 2 (2)
Multiple heart failure symptoms (Cardiac disorders) | 14 (14)
Ventricular Fibrillation (VF) (Cardiac disorders) | 2 (2)
Ventricular Tachycardia (VT)/Monomorphic VT (Cardiac disorders) | 5 (6)
Nonsustained Ventricular Tachycardia (NSVT) (Cardiac disorders) | 4 (4)
Atrial Fibrillation (AF) (Cardiac disorders) | 11 (12)
Sinus tachycardia (Cardiac disorders) | 3 (3)
Atrial Tachycardia/Other SVT (eg AVRT, AVNRT, EAT) (Cardiac disorders) | 2 (2)
Atrial (Type I) Flutter (Cardiac disorders) | 0 (0)
Hypotension/Orthostatic Hypotension (Cardiac disorders) | 4 (4)
Hypertension/Hypertensive Crisis (Cardiac disorders) | 6 (6)
Cardiogenic shock (Cardiac disorders) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 1 (1)
Peripheral vascular disease (Cardiac disorders) | 1 (1)
Syncope (Cardiac disorders) | 1 (1)
Dizziness (Cardiac disorders) | 3 (3)
Chest pain - Ischemic (Cardiac disorders) | 1 (1)
Chest pain - Other (Cardiac disorders) | 7 (7)
Palpitations (Cardiac disorders) | 1 (1)
Adverse reaction - Hypotension (Vascular disorders) | 2 (2)
Adverse reaction - Anesthesia (Injury, poisoning and procedural complications) | 0 (0)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0)
Adverse reaction - Medication (Injury, poisoning and procedural complications) | 3 (3)
Systemic infection (Blood and lymphatic system disorders) | 0 (0)
Physical trauma (Skin and subcutaneous tissue disorders) | 1 (1)
Abnormal laboratory values (Blood and lymphatic system disorders) | 1 (1)
Localized Infection (Skin and subcutaneous tissue disorders) | 0 (0)
Neurological (Nervous system disorders) | 0 (0)
Gastrointestinal (Gastrointestinal disorders) | 3 (3)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Genitourinary (Reproductive system and breast disorders) | 1 (1)
Renal (Renal and urinary disorders) | 0 (0)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1)
Psychological (Psychiatric disorders) | 0 (0)
Endocrine (Endocrine disorders) | 2 (2)
Cancer (General disorders) | 0 (0)
Multi-system failure (General disorders) | 0 (0)
Elevated threshold - LV PG System (Product Issues) | 1 (1)
Psychological effect due to device therapy - PG System - Subject related (Psychiatric disorders) | 1 (1)
pain at device site (Product Issues) | 1 (1)
Conductor coil fracture - RA Lead (Product Issues) | 1 (1)
Extracardiac stimulation - RV Lead (Product Issues) | 1 (1)
Syncope - Heart failure (Cardiac disorders) | 1 (1)
Hypertension - Heart failure (Cardiac disorders) | 2 (3)
Premature Ventricular Contractions (PVC) (Cardiac disorders) | 1 (1)
Distal thromboemboli (Vascular disorders) | 1 (1)
Pericardial effusion - Unrelated (non study) procedure or device (Cardiac disorders) | 1 (1)
Hematological (Blood and lymphatic system disorders) | 1 (1)
HEENT (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-11): https://cdn.clinicaltrials.gov/large-docs/81/NCT02652481/Prot_SAP_000.pdf